CLINICAL TRIAL: NCT06695156
Title: Exploring the Effect of the Transcendental Meditation® Technique on Migraine Frequency and Functionality: A Single Arm Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi International University (Other)
Responsible Party: Principal Investigator, Fred Travis, Director, Brain Center and PhD Chair of the Department of Maharishi Vedic Science at Maharishi University of Management, Maharishi International University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIU002
Record Dates: First submitted 2024-11-02; First posted 2024-11-19 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-08

CONDITIONS: Migraine; Migraine With or Without Aura
Keywords: Migraine; Meditation; Transcendental Meditation
MeSH Terms: conditions — Migraine Disorders | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: It is a pilot study investigating the impact of Transcendental Meditation on migraine as a basis for a larger randomized control study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exploring the Effect of the Transcendental Meditation® Technique on Migraine (Experimental)
  Interventions: Behavioral: Meditation

INTERVENTIONS:
Behavioral: Meditation — The objective of this study is to assess the safety, feasibility, and effects of the practice of the Transcendental Meditation technique in adults with migraines. This study will involve 30 male and female participants recruited from migraine treatment facilities and migraine support groups in the US. The study will span three months, with all participants practicing Transcendental Meditation (TM) while continuing their usual lifestyle and medication regimen. Pre-data will be collected through symptom analysis, headache patterns, and evaluation questionnaires. All potential subjects will use a migraine App for 30 days prior to inclusion in the study, both as a means of assessing migraine status and of ability to adhere to study protocols during the study. In addition, all subjects will take the PHQ-9 to screen for levels of depression that might impair participation in the study. All the subjects will receive TM instruction, followed by bi-weekly

SUMMARY:
This research will explore the effect of the Transcendental Meditation® Technique on migraine intensity and frequency. It will be a single-arm pilot study involving 30 participants recruited from migraine treatment facilities and support groups in the US.

DETAILED DESCRIPTION:
The objective of this study is to assess the safety, feasibility, and effects of the practice of the Transcendental Meditation technique in adults with migraines. This study will involve 30 participants recruited from migraine treatment facilities and migraine support groups in the US. The study will span three months, with all participants practicing Transcendental Meditation (TM) while continuing their usual lifestyle and medication regimen. Pre-data will be collected through symptom analysis, headache patterns, and evaluation questionnaires. All potential subjects will keep a daily migraine diary for 30 days before inclusion in the study, both to assess migraine status and to adhere to study protocols during the study. All the subjects will receive TM instruction, followed by bi-weekly group meetings and one-on-one sessions for 3 months to monitor progress and ensure correct practice.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of migraine with or without aura, based on ICHD3 criteria
* 6-14 migraine days/month.
* ≥ one-year history of migraines starting before the age of 50.
* ≥ 18 years old or ≤ 60 Years old
* Willing to attend follow-up sessions.
* Willing to practice TM twice a day for 20 minutes.
* Fluent in English.

Willing to continue the same medication without any additional medicine

In good general health, with no other diseases expected to interfere with the study.

Exclusion criteria:

* > 60 years old or < 18 Years old
* Already practicing Transcendental Meditation.
* Pre-diagnosed major systemic illness or unstable medical/psychiatric condition (eg, suicide risk) requiring immediate treatment or that could compromise protocol adherence
* Medication overuse headache (MOH)
* Current/planned pregnancy or breastfeeding
* New prophylactic migraine medicine started within 4 weeks of the screening visit
* Unwilling to maintain stable migraine medication dosages
* Failure to complete baseline headache logs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Frequency and functionality | 6 Months
  Frequency and functionality will be measured by the data recorded in the migraine App.
The Migraine Disability Assessment (MIDAS) to measure frequency and functionality. | 6 Months
Migraine Specific Quality of Life Questionnaire (MSQ), version 2.1 to measure impact on Quality of Life | 6 Months
Questionnaire (MSQ), version 2.1 to measure impact on functionality. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Fred T Travis, PhD, Study Chair — Maharishi International University
Locations (1):
- Georgetown Headache Center and DC area, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is a pilot study, and data will be used to design a larger RCT study.

REFERENCES:
- See also: Migraines and Meditation We are conducting research to see the effect of Transcendental Meditation (TM) on the intensity and frequency of migraines. — https://ashashristi.wixsite.com/migrainestudy